CLINICAL TRIAL: NCT00627471
Title: A 24 Weeks, Randomized, 2 Arms, Controlled, Multi-centre, National, Open-labeled, Parallel Study in Insulin naïve Patients With Type 2 Diabetes to Compare a Lantus Titration Algorithm vs. Physician's Standard Practice
Brief Title: Type 2 Diabetes Management With Lantus® (Malbec: Manejo Con Lantus® de Diabéticos Tipo 2)
Acronym: Malbec
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment in spite of strategies implemented
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_02936
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): This group must follow a defined algorithm. Only the physicians assigned to this group will know the algorithm.
  Interventions: Drug: Insulin Glargine
- B (Active Comparator): This is the control group, following the physician's standard practice.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glargine — For the control group (following the physician's standard practice) a minimum of 4 visits to the clinic is required. Insulin titration and concomitant medications will be done at the discretion of the physician. Strips will be distributed among patients in this group, but there will not be a requirement in frequency or type of SMBG.
  Arms: B
Drug: Insulin Glargine — In the group following the algorithm, fasting SMBG will be asked 3 times a week until FBG<100 mg/dl is achieved. Afterwards, 1 fasting SMBG will be asked weekly. Pre-prandial SMBG will be performed at the discretion of the physician.
  For the group following the algorithm, during the titration period, weekly telephone contacts will be required and a minimum of 4 visits to the clinic.
  Arms: A

SUMMARY:
To compare in terms of HbA1c insulin naive patients with Type 2 Diabetes starting with insulin glargine on an algorithm with insulin naive patients starting with insulin glargine on the physician's standard practice.

To compare in terms of FBG insulin naïve patients starting with insulin glargine on an algorithm with insulin naïve patients starting with insulin glargine on the physician's standard practice.

To compare the percentage of patients achieving HbA1c< 7% in each treatment group.

To compare hypoglycaemic events (minor, severe and nocturnal) between groups.

To compare average insulin dose between groups.

To compare PRO (patients' reported outcomes) between groups.

To compare mean changes in body weight between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes.
* Patients in treatment with OADs (one or more) for at least 1 year who failed metabolic control (HbA1c > 8% and < 11%).
* FBG > 130 mg/dl and < 240 mg/dl.
* BMI < 40 kg/m2 and >25 kg/m2.
* Ability and willingness to follow a tight anti-diabetic therapy and to perform SMBG controls.

Exclusion Criteria:

* C peptide < 0.30 nmol/l.
* Unexplained weight loss of more than 10% of body weight in the last 6 months.
* Pregnant women or women with the intention of becoming pregnant.
* Women with childbearing potential who will not use contraceptive protection.
* Breastfeeding women.
* Patients using or that have used rapid or ultra-rapid acting insulins; except for those patients that have used rapid or ultra-rapid insulins during intercurrences such as AMI, severe infection or surgery.
* Renal impairment defined as serum creatinine >1.4 mg/dl in women and >1.5 mg/dl in men.
* Hepatic impairment defined as GPT or GOT above 2x the normal threshold.
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol (non selective beta blockers and systemic corticosteroids).
* History of drug or alcoholic abuse.
* Diabetic retinopathy with surgical treatment in the 3 months prior to study entry or which may require surgical treatment within 6 months of study entry.
* Clinically relevant cardiovascular, gastrointestinal, hepatic, neurological, endocrine, hematological, oncologic or other major systemic disease making implementation of the protocol or interpretation of the study results difficult, at the discretion of the investigator.
* Evidence of an uncooperative attitude, including poor compliance to any anti- diabetic treatment.
* Known hypersensitivity to insulin glargine.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Mean difference in HbA1c (efficacy) | 6 months

SECONDARY OUTCOMES:
Minor, severe and nocturnal Hypoglycaemic events (safety) | from the begining of the treatment up to 5 days after the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Cristian von Schulz-Hausmann, Study Director — Sanofi-aventis administrative office Argentina
Locations (1):
- Sanofi-aventis administrative office Argentina, Buenos Aires, Argentina